CLINICAL TRIAL: NCT04534062
Title: Effects of PNF D2 Technique With Resistance on Pulmonary Function, Exercise Capacity and Health Status of COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Muhammad Ather Hashmi, Principal Investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAther
Record Dates: First submitted 2020-08-17; First posted 2020-09-01 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: Only participant will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Participants in Group A will perform PNF D2 flexion and extension with free weights (PNF D2 FW) The intensity of exercise will be determined for each individual by using maximum repetition test (1 repetition maximum 1-RM). The intensity will be kept 50 % of the maximal load. 3 sets of PNF D2 FW Flexion (flexion-abduction and external rotation) and PNF D2 FW Extension (extension-adduction-internal rotation) respectively will be performed on each upper limb with 10 repetitions per set. All exercises will be performed with a rest interval of 30 seconds to 1 minute between the sets.
  Interventions: Other: PNF D2 technique
- Group B (Experimental): Participants in this group will perform 3 sets of PNF D2 flexion (flexion-abduction and external rotation) and extension (extension-adduction-internal rotation) respectively with elastic bands after assessing the 1-RM test starting with a lightest resistance and gradually progressing to the higher level. Subsequently, 71% to 86% of 1-RM will be taken as a target range of the resistance for the training that will be applied through Elastic Resistance Band in accordance with values that are provided on the Thera-Band website. Moreover, each set will consist of 10 repetitions for both D2 flexion and Extension and a resting interval of 60 seconds between two consecutive sets. The procedure will be repeated for both limbs.
  Interventions: Other: PNF D2 technique
- Group C (Experimental): The participants in the Group C or control group will perform the PNF D2 flexion and extension without any resistance. Three sets consist of 10 repetitions of each pattern for both upper limbs will be performed with an interval of 60 seconds between two consecutive sets.
  Interventions: Other: PNF D2 technique

INTERVENTIONS:
Other: PNF D2 technique — PNF D2 technique of bilateral upper limb will be performed

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the third leading cause of morbidity and disability with 251 million cases per anum reported worldwide. COPD ranks fourth among the common causes of mortality with an estimated 3 million annual deaths worldwide that is projected to be third by 2020. COPD deaths are more prevalent among the low socio-economic developing countries, estimated up to 90% of the total mortality rate across the globe. In Asia, 13.5% of the total population suffers with COPD. Particularly, in Pakistan every 10th individual suffers with COPD out of which 19.4% are of age above 40 years. Moreover, the problem has been identified as a growing public health concern and a challenge for the clinicians of 21st century. Consequently, the severity of the condition of patients is contributed by exacerbations or co-morbidities, and significant economic burden due to the hospitalizations, absence from work and disability; and its management cost from $1544 to $2335 in Asian countries, annually. However, specific data economic burden for Pakistan is not reported yet. A number of pharmaceutical and non-pharmaceutical treatment options are utilized in the management of COPD; however, pulmonary rehabilitation has been conferred as the corner stone in management of COPD. NICE guidelines emphasize upon the importance of pulmonary rehabilitation for all individuals presenting with COPD; even those who have acutely suffered an exacerbation or underwent recent hospitalization. Moreover, pulmonary rehabilitation consisting of structured exercises regimes and education regarding self-care has been reported to improve COPD symptoms and exercise tolerance; and reduce expenditure of resources on recurrent hospitalization and length of stay. Study has reported that resistance training demonstrated in better improvement in muscular strength than endurance exercise and causes lesser chances of dyspnea while performing activities and is more tolerable than endurance exercise regime. Literature is evident upon that the combination of resistance and endurance training has shown significant improvement in the respiratory parameters. Hence the present study is aimed to incorporate Proprioceptive Neuromuscular Facilitation (PNF) D2 pattern including different types of resistance training in order to determine the response of adjunct therapies on the outcome measures.

DETAILED DESCRIPTION:
Data Collection Procedure:

The participants will be divided into three groups A, B and C on the basis of randomization performed using an envelope technique. The participants in group A will perform PNF D2 with free weights (PNF D2 FW), participants of Group B will perform PNF D2 with elastic bands (PNF D2 ERB) while Group C will be control group and the participants of this group will perform PNF D2 without resistance (PNF D2 WR). Initially, consent will be obtained from all participants after explaining them the protocols of treatment. The Pulmonary Function Test (PFT) will be performed to record pre-intervention spirometric values of FEV1/FVC (Tiffeneau-Pinelli Index), Minute Ventilation (MV), Force expiratory volume in 1 second (FEV1), Forced Vital capacity (FVC), Total Lung Capacity (TLC) and Residual Volume (RV). Similarly, 6 Minute Walk Test (6MWT) and St. George's Respiratory Questionnaire Score will be recorded to determine the exercise capacity and health status score of COPD patient respectively. Following the assessment procedure, both groups will receive 8 weeks of treatment with frequency of 3 sessions per week lasting for 30 minutes approximately.

Intervention Protocol Group A Participants in Group A will perform PNF D2 flexion and extension with free weights (PNF D2 FW) The intensity of exercise will be determined for each individual by using maximum repetition test (1 repetition maximum 1-RM). The intensity will be kept 50 % of the maximal load. 3 sets of PNF D2 FW Flexion (flexion-abduction and external rotation) and PNF D2 FW Extension (extension-adduction-internal rotation) respectively will be performed on each upper limb with 10 repetitions per set. All exercises will be performed with a rest interval of 30 seconds to 1 minute between the sets.

Intervention Protocol Group B Participants in this group will perform 3 sets of PNF D2 flexion (flexion-abduction and external rotation) and extension (extension-adduction-internal rotation) respectively with elastic bands after assessing the 1-RM test starting with a lightest resistance and gradually progressing to the higher level. Subsequently, 71% to 86% of 1-RM will be taken as a target range of the resistance for the training . Moreover, each set will consist of 10 repetitions for both D2 flexion and Extension and a resting interval of 60 seconds between two consecutive sets. The procedure will be repeated for both limbs.

Intervention Protocol Group C The participants in the Group C or control group will perform the PNF D2 flexion and extension without any resistance. Three sets consist of 10 repetitions of each pattern for both upper limbs will be performed with an interval of 60 seconds between two consecutive sets.

After 8 weeks of training, the pulmonary function test (PFT), 6 Minute Walk Test and George's Respiratory Questionnaire scores will be recorded for post intervention readings. Results will be recorded and statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed COPD patients of Age 40 and above (Razzaq et al., 2018)
* COPD grade 2 and 3 according to GOLD classification (Berry et al., 2018) (Goldcopd.org, 2019)
* COPD patient both male and female

Exclusion Criteria:

* Individuals with either fractures of ribs or upper limb
* Pulmonary Effusion,
* Pulmonary Edema,
* Embolism,
* Pneumothorax
* Hemothorax

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-22 (Estimated); Study Completion 2021-02-22 (Estimated)

PRIMARY OUTCOMES:
FEV1/FVC Ratio(Pre-intervention) | Baseline
  Spirometry is used to assessed the FEV1/FVC (Forced Expiratory Volume in 1st second/ Forced Vital Capacity) Ratio
FEV1/FVC Ratio(Pre-intervention) | On the completion of 8 weeks of intervention
  Spirometry is used to assessed the FEV1/FVC (Forced Expiratory Volume in 1st second/ Forced Vital Capacity) Ratio
FVC (Forced Vital Capacity) (Pre-intervetion) | Baseline
  Spirometry is used to assessed Forced Vital Capacity
FVC (Forced Vital Capacity) (Pre-intervetion) | On the completion of 8 weeks of intervention
  Spirometry is used to assessed Forced Vital Capacity
Exercise Capacity | Baseline
  6 minute walk test is used to assessed the exercise capacity
Exercise Capacity | On the completion of 8 weeks of intervention
  6 minute walk test is used to assessed the exercise capacity
Health Status | Baseline
  St. George Respiratory Questionnaire is used to assessed the health status
Health Status | On the completion of 8 weeks of intervention
  6 minute walk test is used to assessed the exercise capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No